CLINICAL TRIAL: NCT05877391
Title: A Novel Intervention to Improve Care for Older Sexual and Gender Minority (SGM) Adults With Serious Illness and Especially Those With Alzheimer's Disease and Related Dementias (ADRD)
Brief Title: Intervention to Collect and Utilize Sexual Orientation and Gender Identity (SOGI) Information in Hospice
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 212337
Record Dates: First submitted 2023-03-30; First posted 2023-05-26 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Sexual and Gender Minorities; Hospice; Alzheimer's Disease and Related Dementias
MeSH Terms: conditions — Coitus; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SGM Communication Intervention (Other): The goal of the arm is to train hospice staff in person-centered communication that includes SOGI data collection to promote authentic end-of-life care for SGM patients and their caregivers.
  Interventions: Behavioral: SGM Communication Intervention

INTERVENTIONS:
Behavioral: SGM Communication Intervention — Evaluate the feasibility and acceptability of the SGM communication intervention by hospice staff. I will pilot test the training with hospice staff to refine the content and delivery of the training. Outcomes in the pilot clinical trial will include feasibility, acceptability, and staff satisfaction with training.

SUMMARY:
Older sexual and gender minority (SGM) patients are at risk for receiving inequitable end-of-life care; those with Alzheimer's disease and related dementias (ADRD) are at particularly high risk. Failure to collect and integrate sexual orientation and gender identity (SOGI) data to identify patients' informal support systems may have adverse health consequences for SGM older adults, particularly for those dependent on informal caregivers to provide in-home support and assist with activities of daily living. The goal of this K01 is develop a novel training for hospice staff in person-centered communication that includes SOGI data collection to promote authentic end-of-life care for SGM patients and their caregivers.

DETAILED DESCRIPTION:
Collecting representative and inclusive data about sexual orientation and gender identity (SOGI) is a critical component of combating the devastating health disparities affecting sexual and gender minority (SGM) older adults. This is particularly crucial for patients living with ADRD, which is widely regarded as a family disease requiring the active caregiver involvement, particularly with advanced disease. Failure to collect and integrate SOGI data to identify patients' informal support systems may have adverse health consequences for SGM older adults, particularly for those dependent on informal caregivers to provide in-home support and assist with activities of daily living. Improper identification of chosen family and caregivers contributes to incomplete care delivery and disenfranchised grief. Given the historical discrimination experienced by older SGM people, adding SOGI questions without proper training has the potential to harm patients and create staff discomfort rather than foster inclusive interactions. For this career development award, I propose to characterize SOGI data collection challenges from patients and caregivers enrolling in hospice while exploring understudied intersections, such as SGM people living with ADRD, and how they affect staff approaches to delivering person-centered care. These insights will be used to develop and pilot test an intervention to train hospice interdisciplinary team (IDT) staff to sensitively collect and utilize SOGI data to improve communication with SGM patients and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* 18 years and above

Exclusion Criteria:

--People under 18, pregnant women, prisoners, and people who are decisionally challenged will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Barriers and facilitators to communicating with SGM older adults and perceptions and preferences for asking/disclosing SOGI | Years 1-2
  Evaluating barriers and facilitators to creating an affirming environment where SGM patients and their caregiver feel included and safe to disclose; perceptions and preferences for asking for/disclosing SOGI.
Content of training | Years 2-3
  Iteratively develop content areas with a focus on facilitating conversations with patients who are different than you.
Delivery of content | Year 3-4
  Determine acceptable, replicable, and scalability of content.
Feasibility and assessment of training | Year 5
  Evaluate feasibility of training intervention through simulation with standardized patients and hospice staff. Including evaluating content and delivery of the training and assess delivery of training, feasibility, comfort and confidence the training, incorporation into practice, and evaluation of content.

SECONDARY OUTCOMES:
Sources of bias and stigma | Years 1-2
  Identify sources of stigma (anticipated, internalized, and experienced) and sources of bias (e.g. community, hospice staff, culture, policies).
Ongoing engagement around SOGI-informed care | Years 2-3
  Evaluate means for ongoing engagement of the SGM community for ongoing, authentic, training delivery.
Accessibility | Years 3-5
  Evaluate accessibility of training intervention ussing simulation with standardized patients and hospice staff, pilot test the training to refine the content and delivery of the training and assess accessibility and satisfaction with training.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Aurora, Colorado, United States